CLINICAL TRIAL: NCT04320173
Title: An Open Label, Three-period, Single-application, Adhesion Performance Study ZTlido® (Lidocaine Topical System) 1.8% Compared to Lidoderm® (Lidocaine Patch 5%) and Versatis® (Lidocaine Medicated Plaster 5%) in Healthy, Adult, Human Subjects
Brief Title: Adhesion Performance Study of Lidocaine Topical System 1.8% Compared to Lidocaine Patch 5% and Lidocaine Medicated Plaster 5% in Healthy, Adult, Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scilex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SCI-LIDO-ADH-002
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Healthy
MeSH Terms: interventions — Lidocaine; Lidoderm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lidocaine Patch (Sequence ABC) (Experimental): Subjects received all three topical lidocaine products in Periods 1, 2, and 3. The sequence in which they received the lidocaine products was determined by random assignment. For subjects in Arm 1, 3 lidocaine 1.8% patches were applied in Period 1, and 3 lidocaine 5% patches were applied in Period 2, and 3 lidocaine 5% medicated plasters were applied in Period 3.
  Interventions: Drug: Lidocaine patch 1.8%; Drug: Lidocaine patch 5%; Drug: Lidocaine medicated plaster 5%
- Lidocaine Patch (Sequence CAB) (Experimental): Subjects received all three topical lidocaine products in Periods 1, 2, and 3. The sequence in which they received the lidocaine products was determined by random assignment. For subjects in Arm 2, 3 lidocaine 5% medicated plasters were applied in Period 1, and 3 lidocaine 1.8% patches were applied in Period 2, and 3 lidocaine 5% patches were applied in Period 3.
  Interventions: Drug: Lidocaine patch 1.8%; Drug: Lidocaine patch 5%; Drug: Lidocaine medicated plaster 5%
- Lidocaine Patch (Sequences BCA) (Experimental): Subjects received all three topical lidocaine products in Periods 1, 2, and 3. The sequence in which they received the lidocaine products was determined by random assignment. For subjects in Arm 3, 3 lidocaine 5% patches were applied in Period 1, and 3 lidocaine 5% medicated plasters were applied in Period 2, and 3 lidocaine 1.8% patches were applied in Period 3.
  Interventions: Drug: Lidocaine patch 1.8%; Drug: Lidocaine patch 5%; Drug: Lidocaine medicated plaster 5%

INTERVENTIONS:
Drug: Lidocaine patch 1.8% — Three patches are applied to the subject's back for 12 hours.
  Other Names: Lidocaine topical system 1.8%; ZTlido
Drug: Lidocaine patch 5% — Three patches are applied to the subject's back for 12 hours.
  Other Names: Lidoderm
Drug: Lidocaine medicated plaster 5% — Three plasters are applied to the subject's back for 12 hours.
  Other Names: Versatis

SUMMARY:
The primary objective of this study was to evaluate the adhesion performance of ZTlido® (lidocaine topical system) 1.8% compared to adhesion performance for Lidoderm® (lidocaine patch 5%) and Versatis® (lidocaine medicated plaster 5%).

ELIGIBILITY:
Key Inclusion Criteria:

* Must be healthy based on by medical history, laboratory work, and physical exam with BMI range between 18.00 and 30.00 kg/m2 inclusive.
* Non-smokers
* Be at least 18 years of age
* If childbearing potential, use of acceptable form of birth control
* In the case of females of childbearing potential, have a negative serum pregnancy test

Key Exclusion Criteria:

* Allergy or known hypersensitivity to lidocaine, amide-type local anesthetics, or any component of the product formulation
* Any major medical illness 3 months prior or any significant history or ongoing chronic medical illness
* Presence of any current dermatological condition including psoriasis, eczema, and atopic dermatitis
* Presence of any skin condition such as scratches, cuts, scars, abrasions, excessive hair, tattoos, moles, recently shaved skin, uneven skin texture, irritated (e.g., redness, rash or having blister, etc.) or excessively oily skin at the application areas that may affect the application of the product or adhesion properties of the product.
* History of significant dermatologic cancers (e.g., melanoma, squamous cell carcinoma) except basal cell carcinomas that were superficial and do not involve the investigative site
* History of addiction, abuse, and misuse of any drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-22 (Actual)

PRIMARY OUTCOMES:
Mean Adhesion Score (FDA scale) | 12 hours post-dose
  Adhesion of the product to the skin is assessed by the FDA 0-4 scoring system. The scoring for adhesion is indicated as follows: 0 = ≥ 90% Adhered (essentially no lift off the skin), 1 = ≥ 75% to < 90% Adhered (some edges only lifting off the skin), 2 = ≥ 50% to < 75% Adhered (less than half of the patch lifting off the skin), > 0% to < 50% Adhered but not detached (more than half of the patch lifting off the skin without falling off), and 4 = 0% adhered (patched completely detached). Adhesion is assessed every 3 hours for 12 hours. The mean cumulative adhesion score is calculated as the sum of scores at each assessment time point divided by the total number of observations.
Mean Adhesion Score (EMA scale) | 12 hours post-dose
  Adhesion of the product to the skin is assessed by the EMA 0-6 scoring system. The scoring for adhesion is indicated as follows: 0 = < 70% Adhered, 1 = > 70% Adhered, 2 = > 75% Adhered, 3 = > 80% Adhered, 4 = > 85% Adhered, 5 = > 90% adhered, and 6 = > 95% Adhered. Adhesion is assessed every 3 hours for 12 hours. The mean cumulative adhesion score is calculated as the sum of scores at each assessment time point divided by the total number of observations.

SECONDARY OUTCOMES:
Dermal Response Score | 12.5 and 14 hours post-dose
  Product tolerability is assessed by Dermal Response Score. The application site is evaluated 30 minutes and 2 hours after product removal (12.5 and 14 hours post-dose, respectively). Response score from 0 to 7; 0= No evidence of irritation, 1= Minimal erythema, barely perceptible, 2= Definite erythema, readily visible; minimal edema or minimal papular response, 3= Erythema and papules, 4= Definite edema, 5= Erythema, edema and papules, 6= Vesicular eruption, 7= Strong reaction spreading beyond test (i.e., application) site.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip LaStella, MD, Principal Investigator — TKL Research, Inc.
Locations (1):
- TKL Research, Inc., Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Gudin J, Webster LR, Greuber E, Vought K, Patel K, Kuritzky L. Open-Label Adhesion Performance Studies of a New Lidocaine Topical System 1.8% versus Lidocaine Patches 5% and Lidocaine Medicated Plaster 5% in Healthy Subjects. J Pain Res. 2021 Feb 23;14:513-526. doi: 10.2147/JPR.S287153. eCollection 2021. PMID 33654425